CLINICAL TRIAL: NCT02361541
Title: Determination of Hepatitis C Prevalence, Genetic Diversity and Treatment Eligibility in an HIV Patient Cohort in Phnom Penh, Cambodia
Brief Title: Determination of HCV Prevalence in a HIV Patient Cohort in Phnom Penh, Cambodia
Acronym: HCV-Epi
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Sihanouk Hospital Center of HOPE (SHCH), Phnom Penh, Cambodia (Unknown); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-Epi
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Left over biological samples (whole blood plasma and serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV screening: All adult patients of an existing HIV cohort
  Interventions: Procedure: HCV screening

INTERVENTIONS:
Procedure: HCV screening — HCV antibody screening, liver function tests, full blood count and HbsAg will performed. Additional blood samples will be taken for further HCV diagnostic work-out (polymerase chain reaction (PCR) and genotyping). For patients with current HCV infection, liver ultrasound, transient elastography - Firbroscan and further lab analysis will be performed.

SUMMARY:
Hepatitis C (HCV) is an important global public health problem, disproportionately affecting HIV positive populations. Asia and Africa account for most of the co-infection burden, but access to HCV screening and treatment is still very limited. It is expected though, with the recent therapeutic advances and increasing global advocacy efforts, that HCV treatment should become a feasible option in the near future.

Sihanouk Hospital Center of HOPE (Phnom Penh, Cambodia) is catering for one of the largest HIV cohorts of the country, followed in an ambulatory settings. In this cohort, the prevalence of HCV co-infection will be determined, as well as HCV genotype diversity and the severity of liver disease. The researcher will also explore the performance of simple blood tests/panels as predictors of significant fibrosis and/or cirrhosis.

Patients will attend two study-visits. All adult patients of the HIV patient cohort of SHCH will be proposed HCV testing during their next HIV follow-up consultation, following the latest algorithm of the Centre for Disease Control (CDC) (May 2013). Anamnesis and clinical examination will focus, additionally to routine practice, on presence of general and HCV liver-disease related features. Laboratory analyses will include basic HIV tests (CD4), and tests for liver function such as Hepatitis B surface antigen (HbsAg) .

During the following routine HIV follow-up consultation, the results of HCV testing will be explained to the patient. If the patient is HCV negative, his/her study participation ends here. If currently infected with HCV, the clinician will repeat the HCV liver-disease (extra-hepatic & hepatic) related anamnesis and clinical examination, and prescribe additional blood tests for the non-invasive liver fibrosis/cirrhosis blood panel tests, liver and kidney function. Patients will moreover be asked to undergo a liver ultrasound and liver stiffness measurements.

DETAILED DESCRIPTION:
Hepatitis C (HCV) is an important global public health problem, disproportionally affecting HIV positive populations. Asia and Africa account for most of the co-infection burden, but access to HCV screening and treatment is still very limited. The high cost and complexity of current diagnostic and treatment algorithms are major bottlenecks and the linked lack of accurate HCV prevalence estimates and treatment-need data do not allow for robust treatment advocacy and program planning. Cambodia is not an exception.

It is expected though, with the recent therapeutic advances and increasing global advocacy efforts, that HCV treatment should become a feasible option in the near future. Sihanouk Hospital Center of HOPE (Phnom Penh, Cambodia) is catering for one of the largest HIV cohorts of the country, and it is planning to engage in HCV treatment from 2014 2015 onwards, with a double objective of direct patient benefit and catalyst role at national level, as in the past when starting its antiretroviral (ARV) program.

Within this specific setting, the researchers plan to determine the prevalence of HCV co-infection, HCV genotype diversity and severity of liver disease in this HIV patient cohort, followed in an ambulatory setting. The researchers will also explore the performance of simple blood tests/panels as predictors of significant fibrosis and/or cirrhosis .

The current HCV diagnostic procedures (and tools), as applied in this study, are too expensive and resource-demanding to allow for scalability in resource limited settings. Thus, the researchers plan to set up during this study a biobank with samples of a clinically well described HIV patient population. These samples should allow constituting a well-balanced panel for evaluation of future 'more scalable' HCV diagnostic tools.

Patients will attend two study-visits. All adult patients of the HIV cohort will be proposed HCV testing during their next regular HIV follow-up consultation. HCV testing will follow the latest algorithm of the Centre for Disease Control (CDC) (May 2013). During this same consultation, anamnesis and clinical examination will focus, additionally to routine practice ,on presence of general and HCV liver-disease related features. Laboratory analyses will also include basic HIV (CD4), and tests for liver function such as Hepatitis B surface antigen (HbsAg).

During the following routine HIV follow-up consultation (2-3 months later), the results of HCV testing will be explained to the patient. If the patient is HCV negative, his/her study participation ends here. If currently infected with Hepatitis C, the clinician will repeat the HCV liver-disease (extra-hepatic & hepatic) related anamnesis and clinical examination and prescribe additional blood tests for the non-invasive liver fibrosis/cirrhosis blood panel tests, liver and kidney function. Patients will moreover be asked to undergo a liver ultrasound and liver stiffness measurements.

The biobank will be set up with left over biological samples (whole blood plasma and serum) and comprehensive clinical information of all patients who give additional consent for this scope. Both biological samples and clinical information will be coded, to ensure confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> or = 18 years old)
* Documented HIV positive
* In regular HIV care follow-up (min. 2 consultations in the last six months prior to the study)
* Willing and able to provide written informed consent

Exclusion Criteria:

• HIV patients with currently taking Hepatitis C treatment or with a history of prior hepatitis C treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients in a cohort of HIV-positive patients in Cambodia
Sampling Method: Non-Probability Sample
Enrollment: 3045 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of HCV infection | Baseline
  Seroprevalence of HCV infection in the HIV patient cohort

SECONDARY OUTCOMES:
Proportion of current HCV infection | Baseline
  Proportion of currently infected with HCV among the HCV-IgG positive HIV patients
Proportion of HCV false-positives | Baseline
  Proportion of HCV biologically false-positives among HCV-IgG positive screening
HCV genotypes | Baseline
  Proportions of different HCV genotypes
Severity of liver disease in HCV patients | Baseline
  To determine the severity of liver disease by transient elastography in this coinfected cohort
HCV diagnostic accuracy | Baseline
  To compare the diagnostic accuracy of commonly available blood panel tests for fibrosis staging in this coinfected cohort, with liver stiffness measurement (considered as reference standard).

CONTACTS AND LOCATIONS:
Overall Officials: Anja De Weggheleire, MD, Study Director — Institute of Tropical Medicine, Antwerp, Belgium; An Sokkab, MD, Principal Investigator — Sihanouk Hospital Center of HOPE (SHCH), Cambodia
Locations (1):
- Sihanouk Hospital Center of HOPE (SHCH), Cambodia, Phnom Penh, Cambodia

REFERENCES:
- [Derived] De Weggheleire A, De Baetselier I, An S, Goletti S, Suin V, Thai S, Francque S, Crucitti T, Lynen L, Van Gucht S, Kabamba BM. Challenges to Differentiate Hepatitis C Genotype 1 and 6: Results from A Field-Study in Cambodia. Infect Dis Ther. 2020 Sep;9(3):657-667. doi: 10.1007/s40121-020-00304-7. Epub 2020 May 30. PMID 32474893